CLINICAL TRIAL: NCT03848897
Title: Immersive Virtual Reality Using a Head Mounted Display and Modelling Using Machine Learning Algorithms to Assess Risk of Falling in the Elderly and Patients With Parkinson's Disease.
Brief Title: Contribution of Virtual Reality and Modelling in Falling Risk Assessment in Elderly and Parkinson's Disease Patients
Acronym: PrévSim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: OHS - Office d'Hygiène Sociale (Unknown); ONPA - Office Nancéien des Personnes Agées (Unknown); University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-A02637-48
Record Dates: First submitted 2019-01-30; First posted 2019-02-21 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Aging Disorder; Parkinson Disease
Keywords: Virtual reality; Human metrology; Motor behavior; Modeling; Ageing; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non falling elderly (Experimental)
  Interventions: Other: Metrology of motor behavior
- Falling elderly (Experimental)
  Interventions: Other: Metrology of motor behavior
- Non falling patients with Parkinson's disease (Experimental)
  Interventions: Other: Metrology of motor behavior

INTERVENTIONS:
Other: Metrology of motor behavior — Biomechanical, physiological, psychological and behavioral analyses

SUMMARY:
The process of ageing affects at the same time the sensory, cognitive and driving functions. Furthermore, ageing is often accompanied by pathologies increasing the effects of the senescence. An ageing subject will have then more difficulties in maintaining balance control and will have a falling risk with sometimes critical consequences for the quality of life.

The risk of fall is estimated by tests at the same time of current life and with scores of sensitivity and specificity which must be improved. In a review including 25 studies (2 314 subjects), show a sensitivity of 32 % and a specificity of 73 % on the test "Timed Up and Go" (TUG) with a threshold at 13.5 seconds.

In addition, the fall occurs in a multifactorial context when a subject interacts with his environment. It therefore seems essential to test balance control or falling risk of individuals as close as possible to the situations of daily life. This research, based on the TUG, will aim to assess the neuro-psycho-motor behavior of subjects in situations close to daily life using a Virtual Reality (VR) and Human Metrology platform.

The results could ultimately lead to increased sensitivity and specificity in assessing the risk of falling with a TUG performed in VR, compared to the classic TUG, which is commonly used by healthcare professionals and thus allow for earlier or more appropriate management of the subject in preventing the risk of falling. This could allow healthcare professionals to better understand the risk of falling and thus guide medical recommendations and prescribing, particularly in terms of appropriate physical activity programs.

ELIGIBILITY:
Inclusion Criteria:

Non-faller elderly

* Male and female
* Age between 65 and 80 years old
* Autonomous
* Reporting no fall in the last 12 months

Fallers elderly

* Male and female
* Age between 65 and 80 years old
* Autonomous
* Reporting at least 1 fall in the last 12 months

Non-faller Patients with Parkinson's disease

* Male and female
* Age between 65 and 80 years old
* Autonomous
* Reporting no fall in the last 12 months
* Dopa-sensitive
* In ON period of treatment of Parkinson's disease

Exclusion Criteria:

* Hearing loss preventing understanding of the instructions and listening to the sound message
* Visual acuity not compatible with the test procedure in virtual reality
* Inability to move without assistance
* Not understanding written and oral French, illiteracy, dementia
* Treatment including psychotropic drugs
* Person in emergency situation,
* Major person subject to a legal protection measure (guardianship, curator, safeguard of justice),
* Major person unable to express his consent,
* Hospitalized person,
* Person deprived of liberty by a judicial or administrative decision, the persons being the object of psychiatric care by virtue of articles L. 3212-1 and L. 3213-1 of the french Code of Public Health,
* Person likely, in the opinion of the investigator, not to be cooperating or respectful of the obligations inherent to participation in the study
* Person with a predisposition to epilepsy

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up & Go in virtual reality (VR) | Baseline
  Time

SECONDARY OUTCOMES:
Timed Up & Go (non VR condition) | Baseline
  Time
Validation of the TUG in VR condition | 1 year follow-up
  Sensitivity and specificity of the TUG and TUG VR conditions
Correlation between TUG and TUG VR times and fall follow-up | 1 year follow-up
Kinematics analysis | Baseline
  Measurement of full body motion (coordinates on x, y, z axis) in function of the time during the virtual reality tasks
Kinetics analysis | Baseline
  Measurement of plantar pressure evolution (force in Newton) in function of the time during the virtual reality tasks
Physiological analysis 1 | Baseline
  Measurement of heart pace evolution (bpm) in function of the time during the virtual reality tasks
Physiological analysis 2 | Baseline
  Measurement of breathing evolution (frequence) in function of the time during the virtual reality tasks
Physiological analysis 3 | Baseline
  Measurement of galvanic skin response evolution (µSiemens) in function of the time during the virtual reality tasks
Visual attention analysis | Baseline
  Measurement of the gaze focused on virtual objects parameters (number of gazed on each object and time spend focused on the said object)
Psychology analysis 1 | Baseline
  Measurement of the fear of falling (Fall Efficacy Scale-International from Tinetti with a score from 16 to 64)
Psychology analysis 2 | Baseline
  Measurement of the fear of falling (Activities specific Balance Confidence - Scale from Powell & Myers with a score from 0 to 45)
Psychology analysis 3 | Baseline
  Measurement of the coping strategies (Ways of Coping Checklist from Folkman & Lazarus with scores from 1 to 5 for the remembered stress situation subjective evaluation, a score from 10 to 40 for the Problem item, a score from 9 to 36 for the Emotion item and a score from 8 to 32 for the encourgament item).
Automated learning and falling risk estimation | up to 3 years
  Supervised learning with Support Vector Machine, Decision tree, Linear discriminant.
  Using machine learning algorithms is not a measurement but data processing compiling all the data from measurement and comparing them to the number of fall during the year follow up. Machine learning algorithms will learn from these data to classify any new participant into a profile "with a low risk of fall", "with a high risk of fall" or "without a risk of fall".

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No